CLINICAL TRIAL: NCT03076333
Title: Utility of PET/MR in Assessing Response to Neoadjuvant Radiation Therapy in the Treatment of High Grade Sarcomas
Brief Title: PET/MR in Assessing Response to Neoadjuvant Radiation Therapy in the Tx of High Grade Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1615
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-01

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm: PET/MR (Experimental): Each patient will undergo three combined PET/MR scans. The pre-treatment PET, mid-treatment PET and MR, and post-treatment PET are for research purposes and not part of the patient's standard of care (pre-treatment MR and post-treatment MR).
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — Patient will be scheduled for a pre-treatment PET/MR and proceed to neoadjuvant radiation therapy per the direction of the radiation oncologist. At the end of the second week of radiation therapy the patient will undergo a mid-treatment PET/MR. The patient will the complete their radiation therapy. Four weeks after radiation therapy the patient will undergo a post-treatment PET/MR, and proceed for curative intent surgery at 6-8 weeks post radiation if they are still surgical candidates.

SUMMARY:
Purpose: To assess the utility of PET/MR in assessing response to neoadjuvant radiation therapy in the treatment of high grade sarcomas.

Participants: Adult patients with potentially curable high grade sarcomas that are being treated at UNC with neoadjuvant radiation therapy followed by potentially curative surgical resection.

Procedures (methods): Patients who are being treated for potentially curable high grade sarcomas with neoadjuvant radiation therapy followed by surgical resection undergo pre-treatment, mid-treatment, and post-treatment PET/MR and the response to treatment is assessed by evaluating change in size and FDG avidity. Patients then undergo curative intent resection and are followed. Their pathology is reviewed for treatment affect as is assessed by percent necrosis, size, and resection margins. Patients are followed and assessed for recurrence.

DETAILED DESCRIPTION:
Investigators propose that a PET/MR study at the midpoint of radiation treatment will accurately predict which patients will respond to neoadjuvant radiation therapy. The study will enroll patients with high-grade sarcomas as identified by preoperative biopsy that will be treated with neoadjuvant radiation into the study. The standard of care for these patients is to receive MRI scans at pre-treatment and post-treatment time points. Patients in this study will receive their standard pre- and post-treatment imaging in the form of PET/MR, with PET conducted simultaneously with MRI, and within the context of the study they will also receive one additional PET/MR at the end of the second week of therapy. These patients will then receive curative intent surgery and be followed in the usual fashion and assessed for local and/or distant recurrent disease. The pathology will be assessed for completeness of resection and percent of necrosis. On the basis of pathology, patients will be classified as responsive or non-responsive to therapy. Quantitative measures from PET and MRI will be computed: the change in PET tumor-mean standardized uptake value (SUV) and tumor size as assessed by MRI, from pre- to post-treatment, and from pre- to mid-treatment. The image-based quantitative measures will be correlated with the pathology outcomes to evaluate predictability of the image measures for treatment response. Patients will be followed with the intent of further correlating image measures with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age (no upper age limit)
* Signed, IRB-approved written informed consent
* Must have a biopsy-proven high-grade retroperitoneal or soft tissue extremity sarcoma confirmed by independent evaluation of a UNC sarcoma specialized pathologist.
* Must have surgically curable disease as evaluated by initial imaging by our UNC surgeons.
* Must be in acceptable health to undergo radiation therapy and curative intent surgery as assessed by UNC surgeons and radiation oncologist.
* Must be able to understand and comply with study procedures for the entire length of the study.
* Must receive their neoadjuvant radiation therapy and curative intent surgery at UNC Hospitals - Chapel Hill location.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to each PET/MRI

Exclusion Criteria:

* Inability to tolerate MRI (e.g., inability to lie flat for >1 hour)
* Presence of pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes or near pelvis that would create excessive imaging artifact
* Poorly controlled diabetes mellitus
* Creatinine > 1.8 mg/dL OR GFR < 30mL/min
* Body Mass Index (BMI) > 35
* Active vaginal bleeding requiring packing and emergent radiation therapy
* Pregnancy or lactating female
* History of a prior malignancy within past 5 years are excluded unless they have been disease free for 3 or more years
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study
* Evidence of distant disease on physical exam or initial imaging
* Medical conditions precluding radiation therapy or curative intent surgery
* Previous radiation exposure precluding radiation therapy
* Had serious reaction to contrast agent
* Incarcerated or otherwise institutionalized at time of enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lalush, PhD, Principal Investigator — UNC Biomedical Engineering
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm: PET/MR
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult patients with potentially curable high grade sarcomas that being treated at UNC with neoadjuvant radiation therapy followed by potentially curative surgical resection were to be recruited.
Arm/Group | Single Arm: PET/MR
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 69 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3
Pre-treatment tumor SUV mean [Mean (Full Range); unit: SUV] | 3.78 [2.43 to 5.12]

OUTCOME MEASURES:

1. Primary Outcome: PET Activity Estimates at Midpoint of Treatment as Compared to Baseline
Description: Primary endpoint is the determination of differences among response groups in PET activity estimates from PET/MR imaging at the midpoint of treatment as compared to baseline. The measure is computed as the change in mean SUV from the baseline PET-MR scan to the scan at the end of the second week of therapy. Treatment response will be determined on final pathological evaluation of the resected specimens in patients who undergo curative intent surgery after neoadjuvant radiation in high grade sarcomas. This will be measured by a single sarcoma specialized pathologist and will be categorized as to the percentage of necrosis, with >90% necrosis considered to be complete response.
Time Frame: At the end of the second week of radiation therapy, a mid-treatment PET/MR is obtained.
Population: All participants
Measure: Mean (Full Range); unit: SUV
Arm/Group | Single Arm: PET/MR
Number analyzed (Participants) | 3
SUV | .44 [-.3 to 2.72]

2. Secondary Outcome: PET Activity Estimates at Endpoint of Treatment as Compared to Baseline
Description: A secondary endpoint is the determination of differences among response groups in PET activity estimates from PET/MR imaging at the endpoint of treatment as compared to baseline. The measure is computed as the change in mean SUV from the baseline PET-MR scan to the scan taken four weeks after completion of therapy.
Time Frame: A post-treatment PET/MR is obtained at 4 weeks post radiation.
Population: All participants
Measure: Mean (Full Range); unit: SUV
Arm/Group | Single Arm: PET/MR
Number analyzed (Participants) | 3
SUV | -.51 [-1.04 to -.03]

ADVERSE EVENTS:
Time Frame: Adverse events collected day of imaging up until time of surgery, an average of 10 weeks.
Arm/Group | Single Arm: PET/MR
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Small numbers of subjects limit data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03076333/Prot_SAP_000.pdf